CLINICAL TRIAL: NCT05045352
Title: Ultrasound Guided Subclavian Vein Cannulation. Echogenic Needles Versus Non-echogenic Needles
Brief Title: Echogenic Versus Non-echogenic Needles for Venous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trine Kåsine, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REK 85090
Record Dates: First submitted 2021-09-03; First posted 2021-09-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Vascular Access Complication
Keywords: vascular access,; ultrasound guided; echogenic needles

STUDY DESIGN:
Intervention Model Description: Two arms Venous access either with echogenic needles or with non-echogenic needles
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be anesthetized and asleep Outcome assessor will not be in the operating theater during the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echogenic needle (Active Comparator): venous access performed under ultrasound guidance with echogenic needles
  Interventions: Device: echogenic needles for intravenous access
- Non-Echogenic needles (No Intervention): venous access performed under ultrasound guidance with non-echogenic needles

INTERVENTIONS:
Device: echogenic needles for intravenous access — echogenic needles for intravenous access (subclavian vein) ultrasound guided procedure
  Arms: Echogenic needle

SUMMARY:
Randomized controlled intervention study comparing echogenic needles with non echogenic needles for ultrasound guided venous access in the subclavian vein.

DETAILED DESCRIPTION:
Patients undergoing certain surgical procedures and patients in intensive care unit require a central venous catheter (CVC) for infusion of medicaments and for monitoring. Central venous access (CVA) can be performed both with a blind technique or an ultrasound guided technique. A common place for CVA is the subclavian vein.

While many guidelines recommend the use of ultrasound for jugular access, there are no explicit recommendations for subclavian CVA For ultrasound guided CVA procedures good needle visualization is important to successfully place the needle and catheter in the correct position.

Echogenic needles can give better needle visualization when performing ultrasound guided CVA procedures. Theoretically, the use of echogenic needles should improve performance time and success rates, and reduce complication rates due to a better needling control.

The investigators will investigate the use of echogenic needles for vascular access.

A prospective randomized controlled trial design will be used. Echogenic needles will be compared with non-echogenic (standard) needles. The main null hypothesis states that there is no difference in access time between the needles.

ELIGIBILITY:
Inclusion Criteria:

undergoing a surgical procedure requiring a CVC Patients must be at least 18 years of age. Patients that have given informed written consent.

-

Exclusion Criteria:

* Patients that do not speak or understand Norwegian language.
* Skin disease or infection affecting the whole-body surface or within the area of examination.
* Patients with untreated coagulopathy
* Known vascular abnormality
* Any reason why, in the opinion of the investigators, the patient should not participate.
* Subject participates in a potentially confounding drug or device trial during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Time from skin puncture of the needle until aspiration of venous blood. | 10 sec - 240 sec
  Time from skin puncture of the needle until aspiration of venous blood in the syringe. Time till venous access

SECONDARY OUTCOMES:
Time from skin puncture until catheter in place | 60 sec - 600 sec
  Time from skin puncture until the catheter in place in the subclavian vein.
Success with venous access in first needling attempt | 60 sec - 600 sec
  Success in first attempt is defined as one skin puncture and directly into the subclavian vein
Number of needling attempts before venous access | 60 sec - 600 sec
  Number of attempts is defined as the counted number of needle attempts intermitted by a needle withdrawal of at least 0.5 cm until aspiration of venous blood.
Number of skin punctures | 60 sec - 600 sec
  Number of skin punctures is defined as the counted number of skin punctures until aspiration of venous blood.
The procedure was aborted | 2 minutes - 20 minutes
  Discontinuation of the procedure or change of site for vascular access
Localization of catheter tip in x-ray | 1 day- 7 days
  Catheter misplacement judged by x-ray. X-ray will be performed after the surgery and a blinded observer will describe the localization of the catheter.
The anaesthetists subjective experience with needle visualization | 3 min- 20 min
  After performing the vascular access the anaesthetists are asked about how they found the visualization of the needle using a Numeric Rating Scale
The anaesthetists subjective experience with the needle placement | 3 minutes - 20 minutes
  After performing the vascular access the anaesthetist is asked how the needle placement was using a Numeric Rating Scale
Incidence of Treatment-Emergent Adverse Events, pneumothorax hematothorax | 1 minutes- 1 day
  Adverse events, including information of the seriousness, treatment needed, resolution and relevant judgment concerning the causal relationship with the investigational devices or procedure will be summarized for safety information
Incidence of delayed Treatment-Emergent Adverse Events pneumothorax, hematothorax | 5 minutes - 1 week
  Adverse device effects, including information of the seriousness, treatment needed, resolution and relevant judgment concerning the causal relationship with the investigational devices or procedure will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Trine Kåsine, MD, Principal Investigator — Department of Anaesthesiology Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No